CLINICAL TRIAL: NCT05274009
Title: Evaluating the Efficacy of Cooling Centres for Limiting Heat Strain in Elderly Adults During Extreme Heat Events
Brief Title: Protective Cooling Measures to Safeguard Elderly People From Dangerous Summer Heat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University Research Chair, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-11-21-7566
Record Dates: First submitted 2022-02-25; First posted 2022-03-10 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Hyperthermia; Heat; Weather; Aging; Type2 Diabetes; Hypertension; Heat Stress
Keywords: Heat wave; Cooling center; Heat strain; Cardiovascular strain; Heat and health protection; Extreme heat events; Thermal comfort
MeSH Terms: conditions — Hyperthermia; Hypertension; Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: Participant will complete 3 simulated extreme heat event exposures in random order: i) no cooling center intervention (control); ii) recommended cooling center intervention (1 x 2-hours of brief air-conditioning); and iii) hybrid cooling center intervention (2 x 1-hour interspersed brief air-conditioning)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be informed of the study interventions before providing informed consent but will be blinded to the specific trial condition at each of the 3 laboratory visits (control, recommended cooling, hybrid cooling). Data will be blinded prior to analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extreme heat event simulation + no cooling (control) (Experimental): Adults aged 60-85 years with or without type 2 diabetes and/or hypertension
  Interventions: Other: No cooling (control)
- Extreme heat event simulation + recommended cooling (Experimental): Adults aged 60-85 years with or without type 2 diabetes and/or hypertension
  Interventions: Other: Recommended cooling
- Extreme heat event simulation + hybrid cooling (Experimental): Adults aged 60-85 years with or without type 2 diabetes and/or hypertension
  Interventions: Other: Hybrid cooling

INTERVENTIONS:
Other: No cooling (control) — Participants are exposed to 35°C, 60% relative humidity for 8 hours.
  Arms: Extreme heat event simulation + no cooling (control)
Other: Recommended cooling — Participants are exposed to 35°C, 60% relative humidity for 3 hours, are then moved to an air-conditioned room for 2 hours (~23°C, ~50% relative humidity), and then return to the heat for a final 3 hours.
  Arms: Extreme heat event simulation + recommended cooling
Other: Hybrid cooling — Participants are exposed to 35°C, 60% relative humidity for 2 hours, are moved to an air-conditioned room for 1 hour (~23°C, ~50% relative humidity), return to the heat for 2 hours, move back to the air-conditioned room for 1 hour, and then return to the heat for a final 2 hours
  Arms: Extreme heat event simulation + hybrid cooling

SUMMARY:
With the increasing incidence and severity of extreme heat events accompanying climate change, there is an urgent need for sustainable cooling strategies to protect heat-vulnerable older adults, who are at increased risk of adverse health events during heat stress. Health agencies including the World Health Organization, the United States Centers for Disease Control and Prevention, and Health Canada currently recommend visiting a cooling centre or other air-conditioned location for 1-3 hours per day during extreme heat events to mitigate hyperthermia and strain on the cardiovascular system and therefore the risk adverse health events. However, our recent trial shows that while brief air-conditioning exposure is effective for reducing body temperature and cardiovascular burden in healthy older adults, the physiological impacts of cooling abate quickly following return to the heat. The purpose of this project is therefore to assess whether shorter but more frequent air-conditioning exposure provides more effective cooling than current recommendations (a single 1-3-hour cooling bout) in older adults with or without common chronic health conditions associated with increased vulnerability to extreme heat. This will be accomplished by evaluating physiological strain in older adults with and without diabetes and/or hypertension exposed for 8 hours to conditions reflective of extreme heat events in temperate, continental climates (35°C, 60% relative humidity). Participants will complete 3 separate simulated heat event exposures: i) a control trial (no cooling throughout the 8-hour heat event); ii) a recommended cooling trial (3 hours of heat exposure followed by 2 hours cooling); and iii) a hybrid cooling trial (2 hours of heat exposure followed by 1 hour cooling, another 2 hours heat exposure followed by 1 hour cooling, and a final 2-hour heat exposure).

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 60-85 years
* Male or female
* Body mass index < 35 kg/m2
* For participants with type 2 diabetes: at least one year lapsed since diagnosis and hemoglobin A1c 6.0-10.5%.
* For participants with hypertension: at least one year lapsed since diagnosis or average resting blood pressure >140 systolic or >90 diastolic

Exclusion Criteria:

* Currently smoking or quit <5 years ago
* Moderate or serious medical conditions (other than Type 2 diabetes or high blood pressure), particularly those known to influence physiological responses to heat exposure (e.g., diagnosed heart disease, neurological disorders)
* Heat adapted due to repeated exposure to hot environments (use sauna, recent travel to hot climates, other)
* For participants with type 2 diabetes: "Brittle" diabetes: unpredictable hypo- & hyperglycemia. Severe cardiovascular autonomic or peripheral neuropathy (guidelines.diabetes.ca/cpg)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Core temperature (peak) | 8-hour heat exposure
  Peak rectal temperature measured during the 8-hour heat exposure.
Core temperature (AUC) | 8-hour heat exposure
  Rectal temperature will be measured continuously throughout each exposure and the area under the curve will be calculated.

SECONDARY OUTCOMES:
Heart rate temperature (peak) | 8-hour heat exposure
  Peak rectal temperature measured during the 8-hour heat exposure.
Heart rate (AUC) | 8-hour heat exposure
  Heart rate will be measured continuously throughout each exposure and the area under the curve will be calculated.
Mean skin temperature | Before and continuously throughout each 8 hour exposure
  Mean skin temperature calculated as a weighted average of skin temperatures at 8 body regions.
Arterial blood pressures | Every hour during the 8-hour heat exposure
  Systolic and diastolic pressures measured in triplicate.
SDNN | Every hour during the 8-hour heat exposure
  Standard deviation of normal-to-normal R-R intervals measured via 3-lead ECG.
RMSSD | Every hour during the 8-hour heat exposure
  Root mean squared standard deviation of normal-to-normal R-R intervals measured via 3-lead ECG.
Rate pressure product | Every hour during the 8-hour heat exposure
  Rate pressure product calculated as systolic blood pressure x heart rate.
Body fluid loss | Every hour during the 8-hour heat exposure
  Body fluid loss calculated as a change in body weight from pre-exposure values (corrected for food intake and deification).
Stand test: 30:15 ratio | Prior to and following the 8-hour heat exposure
  30:15 ratio calculated as the ratio of the RR interval measured after 30 heart beats following standing from a supine position to that measured after 15 heart beats.
Stand test: Systolic response to standing | Prior to and following the 8-hour heat exposure
  Fall in systolic blood pressure after standing from a supine position.
Baroreflex sensitivity | Prior to and following the 8-hour heat exposure
  Baroreflex sensitivity determined during cyclic stand-squat manoeuvres.
Change in plasma volume | Prior to and following the 8-hour heat exposure
  Change in plasma volume calculated from venous blood samples (Dill and Costill technique)

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa; Ronald J Sigal, MD, MPH, Principal Investigator — University of Calgary; Robert D Meade, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be available from Dr. Kenny upon reasonable request and signed access agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After study completion
Access Criteria: Reasonable request and signed access agreement